CLINICAL TRIAL: NCT06735716
Title: Comparison of Procedural and Clinical Outcomes Between Robot Assisted and Conventional Manual Approaches in Patients With Coronary Artery Disease Requiring Percutaneous Coronary Intervention
Brief Title: Comparison of Safety and Efficacy Between the Robot-assisted System AVIAR (MX-02) Procedure and Conventional Manual Procedure in Patients Requiring Percutaneous Coronary Intervention
Acronym: RoboticPCI
Status: Not yet recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: LN Robotics inc. (Unknown)
Responsible Party: Principal Investigator, Tae Oh Kim, Principal Investigator, Asan Medical Center
Other Study IDs: 2024-1271
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Robotic PCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A patient who received PCI procedure using a AVIAR.: After the subject is assigned a registration number, the robot-assisted procedure group will undergo percutaneous coronary intervention (PCI) using the clinical trial medical device 'AVIAR (MX-02)', while the conventional manual procedure group will undergo percutaneous coronary intervention (PCI) according to the standard procedure.
- A patient who received PCI procedure wth conventional manual techniques.: After the subject is assigned a registration number, the robot-assisted procedure group will undergo percutaneous coronary intervention (PCI) using the clinical trial medical device 'AVIAR (MX-02)', while the conventional manual procedure group will undergo percutaneous coronary intervention (PCI) according to the standard procedure.

SUMMARY:
The objective of this study is to compare and evaluate the safety and efficacy of robot-assisted procedures using the positioning catheter control device 'AVIAR (MX-02)' versus conventional manual procedures in patients with Stable angina requiring percutaneous coronary intervention (PCI)

DETAILED DESCRIPTION:
A potential subject who meets the 'general inclusion/exclusion criteria' will be admitted before the procedure, undergo pre-procedure treatment according to the institution's standard procedures, and receive coronary angiography on the day of the procedure under local anesthesia. At this time, the investigator will review the 'coronary angiography inclusion/exclusion criteria', and only subjects who meet all the criteria will be enrolled in the clinical trial.

After the subject is assigned a registration number, the robot-assisted procedure group will undergo percutaneous coronary intervention (PCI) using the clinical trial medical device 'AVIAR (MX-02)', while the conventional manual procedure group will undergo percutaneous coronary intervention (PCI) according to the standard procedure.

After the procedure, the subjects will remain in a supine position for approximately 4 hours in the recovery room or hospital room to ensure absolute stability. During this time, the investigator will observe the puncture site for hemostasis and monitor for any adverse events. Within 2 days after the procedure or prior to discharge, the subjects will undergo safety assessments and evaluations for the occurrence of any adverse events or serious adverse events. Additionally, at the 1-month follow-up, all required follow-up tests will be completed, and if no adverse events have occurred or if any previously occurring adverse events have been resolved, the clinical trial for that particular subject will be concluded. However, if any adverse events remain unresolved and are deemed unrelated to the clinical trial by the investigator, the trial may be terminated for that subject. Please note that the above information is a general description of the procedure and criteria for the clinical trial involving percutaneous coronary intervention using the AVIAR (MX-02) device.

ELIGIBILITY:
Inclusion Criteria:

* * General Inclusion Criteria

  1. Adult women and men who are aged ≥19
  2. Those who are suspected of stable angina and need percutaneous coronary intervention
  3. Those who voluntarily decided to participate in this clinical trial and agreed in writing to the informed consent form
  4. Those who are willing to comply with the protocol.

     * Angiographic Inclusion Criteria
  5. If the target lesion is a single lesion.
  6. If the lesion to be treated by coronary angiography (target lesion) is a native coronary artery lesion that has not been previously treated.
  7. If the diameter of the lesioned vessel to be treated by coronary angiography (target vessel) is between 2.5 mm and 4.5 mm (by visual estimate).
  8. If diameter stenosis of the target vessel ≥50% (by visual estimate)

Exclusion Criteria:

* * General Exclusion Criteria

  1. Those with a left ventricular ejection fraction (LVEF) ≤ 30%
  2. Those who have a history of hypersensitivity to contrast agents such as stainless steel, cobalt-chromium, etc.
  3. Those who cannot stop taking antithrombotic drugs (anticoagulants, antiplatelet drugs)
  4. Those diagnosed with thrombocytopenia, thrombocytosis, neutropenia, or leukopenia
  5. Those who have a history of bleeding diathesis or coagulopathy or who refuse transfusion
  6. Those with a history of stroke (CVA) or transient ischemic attack (TIA) within 4 weeks from the screening date
  7. .Those with a history of active peptic ulcer or upper gastrointestinal bleeding within 24 weeks from the screening date
  8. Those with ST-elevation myocardial infarction (STEMI) (for example, those who started myocardial infarction symptoms within 72 hours from the screening date)
  9. Those with a history of cardiogenic shock or cardiac arrest
  10. Those who underwent coronary artery bypass grafting (CABG)
  11. Those who underwent percutaneous coronary intervention (PCI) within 72 hours from the screening date
  12. Those who had a major adverse coronary event (MACE) or a serious adverse event (SAE) after receiving the percutaneous coronary intervention (PCI) within 4 weeks from the screening date
  13. Those who are scheduled to undergo percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within 4 weeks from the end of this clinical trial
  14. Those diagnosed with renal failure or those who are not suitable for angiography due to severe renal dysfunction (creatine >2.0 mg/dL or eGFR (estimated glomerular filtration rate) <30 ml/min) within one week prior to the date of coronary angiography
  15. Pregnant and breastfeeding women
  16. Women of childbearing potential who plan to become pregnant during this clinical trial
  17. A woman* or spouse who is likely to be pregnant does not agree to use contraception in medically acceptable method of contraception** during the clinical trial
  18. Those who are currently participating in other clinical trials or have experience participating in other clinical trials within 12 weeks from the screening date.However, where at least one or more conditions are satisfied, it could be an exception according to an investigator's discretion
* Participated in the observational study expected no effect on the safety and/or effectiveness evaluation of this trial
* Screening failed before any interventional factor is involved-Participated in academic trials like strategic or medical device comparison 19. Other cases where the investigator determines that participation in a clinical trial is inappropriate ethically or because it may affect the study outcome.

  * Angiographic Exclusion Criteria

    1. Those who require manual or mechanical thrombectomy, rotational atherectomy, directional coronary atherectomy (DCA), etc. in addition to stent placement and balloon dilatation 2. When the two-stent technique is required for the side branch of the target bifurcation lesion.

    3. When the investigator determines that PCI is not suitable because the target lesion hasany of the following characteristics:

    ①he target lesion is a chronic total occlusion (CTO) or total occlusion

    ②An ostial lesion in location

    ③The target vessel has evidence of intraluminal thrombus

    ④Moderate or severe calcification at the target lesion or near the target lesion

    ⑤If PCI cannot be performed for other reasons 4. If the investigator determines that the subject is not suitable for robotic-assisted PCI due to clinical and anatomical reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target number of participants for this clinical trial is a total of 80 patients during study duration . If subjects who meet the "Coronary Angiography Selection/Exclusion Criteria" are eligible to be enrolled in the clinical trial. These subjects will undergo the standard pre-procedural preparations and receive local anesthesia on the day of the procedure. After the subject is assigned a registration number, the robot-assisted procedure group will undergo percutaneous coronary intervention (PCI) using the clinical trial medical device 'AVIAR (MX-02)', while the conventional manual procedure group will undergo percutaneous coronary intervention (PCI) according to the standard procedure.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Success Criteria | 48hours
  If the residual stenosis rate of the lesion is less than 30% after completion of percutaneous coronary intervention using an investigational device If major adverse cardiovascular events (MACE)† have not occurred within 48 hours after the procedure or the time of discharge, whichever comes first
Technical Success Criteria | 48hours
  The stent (or balloon catheter) has successfully reached the target lesion without switching to manual manipulation.
Radiation exposure Patient | 48hours
  Patient Radiation exposure (Gy): The total procedure time is defined as the period from the insertion of the guidewire and guide catheter (introducer sheath) to their removal, during which the radiation exposure (DAP, Air Kerma) and fluoroscopy time are measured on the C-arm.
Radiation exposure Operator | 48hours
  Operator radiation (mSv):It is verified by the radiation exposure measured using the personal electronic dosimeter worn by the operator on the chest and the radiation exposure measured on the procedure table.

SECONDARY OUTCOMES:
TEAE | 1month
  Treatment emergent adverse event, TEAE
MACE | 1month
  Major Adverse Cardiovascular Events) occurring in the study subjects during the clinical trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Oh kim, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided